CLINICAL TRIAL: NCT05931952
Title: Comparative Effects Of Buteyko Breathing Techniques And Papworth Method On Pulmonary Functions And Oxygen Saturation In Asthmatic Patients
Brief Title: Comparative Effects Of Buteyko Breathing Techniques And Papworth Method In Asthmatic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0319
Record Dates: First submitted 2023-06-06; First posted 2023-07-06 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Asthma
Keywords: asthma,; breathing exercises; humans; oxygen saturation,; patients
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buteyko breathing technique (Experimental): Buteyko breathing technique and conventional (chest physiotherapy) treatment for 5 times a week for about 20 minutes in one session for a period of 4 weeks. There are three steps involved in buteyko breathing technique.
  Step 1; control pause breathing test (patient is asked to sit in an upright position and take normal breath. After this, asked the patient to take small breath-in for 2s and out for 3s. Control pause phase should not exceed for >30 seconds).
  Step 2; maximum pause or shallow breathing (patient is asked to place fingers under the nose to monitor inflow of air. 2 or 3 flickers of air is taken in and exhale as slowly as possible).
  Step 3; combine step 1 and 2. Bronchial drainage will be performed as a conventional treatment for 2 to 3 minutes in each segment. During that time, patient is asked to take deep and slow breaths followed by cough to help in clearing mucus.
  Interventions: Other: Buteyko breathing technique
- Papworth method (Experimental): Papworth method and conventional chest physiotherapy (bronchial drainage) treatment. Intervention will be given for a period of 5 sessions per week for 1 month. Duration of each session will be 20 minutes. This technique is performed particularly during remission period that make it feasible for respiratory physiotherapist to integrate this method into activities of daily living. Papworth method has five components including Papworth method ameliorates asthmatic symptoms breathing, education, relaxation, combination of breathing and relaxation exercise and home exercises and also improves quality of life.
  Bronchial drainage will be performed as a conventional treatment for 2 to 3 minutes in each segment. During that time, patient is asked to take deep and slow breaths followed by cough to help in clearing mucus.
  Interventions: Other: Papworth method

INTERVENTIONS:
Other: Buteyko breathing technique — Group A: Buteyko breathing technique and conventional (chest physiotherapy) treatment for 5 times a week for about 20 minutes in one session for a period of 4 weeks. There are three steps involved in buteyko breathing technique.
  Step 1; control pause breathing test (patient is asked to sit in an upright position and take normal breath. After this, asked the patient to take small breath-in for 2s and out for 3s. Control pause phase should not exceed for >30 seconds).
  Step 2; maximum pause or shallow breathing (patient is asked to place fingers under the nose to monitor inflow of air. 2 or 3 flickers of air is taken in and exhale as slowly as possible).
  Step 3; combine step 1 and 2. Bronchial drainage will be performed as a conventional treatment for 2 to 3 minutes in each segment. During that time, patient is asked to take deep and slow breaths followed by cough to help in clearing mucus.
  Arms: Buteyko breathing technique
Other: Papworth method — Papworth method and conventional chest physiotherapy (bronchial drainage) treatment. Intervention will be given for a period of 5 sessions per week for 1 month. Duration of each session will be 20 minutes. This technique is performed particularly during remission period that make it feasible for respiratory physiotherapist to integrate this method into activities of daily living. Papworth method has five components including Papworth method ameliorates asthmatic symptoms breathing, education, relaxation, combination of breathing and relaxation exercise and home exercises and also improves quality of life.
  Bronchial drainage will be performed as a conventional treatment for 2 to 3 minutes in each segment. During that time, patient is asked to take deep and slow breaths followed by cough to help in clearing mucus.
  Arms: Papworth method

SUMMARY:
Asthma is an inflammatory condition which is characterized by coughing, sneezing, and shortness of breath. The ratio of asthma is increasing day by day around the globe. According to an estimate, more than 300 million people are affected from this chronic respiratory disorder throughout the world. The asthma is diagnosis on basis of sign and symptoms as there is no gold standard of evaluating the asthma. There are basically two treatment strategies for asthma involving medical management and physiotherapy treatment. In medical treatment, steroid drugs and bronchodilators are given to asthmatic patients. Now a day, the physiotherapy treatment has gained much importance. There are numerous physiotherapy approaches available for rehabilitating asthma patients such as breathing techniques, yoga, and relaxation exercises. Buteyko technique includes three steps (control pause, shallow breathing and combination of step 1 & 2). While, papworth method includes five steps (breathing, education, relaxation, combination of breathing and relaxation exercise and home exercises). The randomized clinical trials will be conducted for this study and data will be calculated using simple random sampling technique. The study will be carried out in Clinical Private (Farooq Clinic) setting Khushab and THQ Khushab for a period of 10 months after approval from research and ethical committee. Firstly, consent will be taken from the study participants. Screening will be done using WHO Quality of Life Scale questionnaire and asthma control test adult scores. Lung spirometry values (FVC, FEV1, & FEV1/FVC) and oxygen saturation will be evaluated at baseline, 2 weeks, and 4 weeks. Patients will be divided into two groups. Group A & Group B. Buteyko breathing technique will be performed to Group A patients and papworth method will be performed to Group B. Chest physiotherapy will be performed to both groups as a conservative treatment at baseline, 2 weeks, and 4weeks

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed asthmatic patients
* Age group 20-60 years
* Both genders
* Lung function (FEV predicted < 80% & FEV1/FVC < 75%)
* Nighttime awakening 3-4 times/month
* Symptoms > 2 days/week

Exclusion Criteria:

* Unstable asthmatic patients
* Acute upper respiratory infection
* History of radiation
* Taking any oral steroid, mental disorder

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
PFT to assess change | baseline and fourth week
  It is the Pulmonary Function Test and these tests are used to measure lungs functions. These are specifically necessary for diagnosis of respiratory diseases. The data calculated from PFT include Force Vital Capacity (FVC), Force Expiratory Volume at 1 second (FEV1), and FEV1/FVC
Asthma Control Test Adult (ACT) to assess change | baseline and fourth week
  Asthma Control Test (ACT) is a clinical tool for evaluation of symptoms of asthmatic patients. It is a 5-item questionnaire for the assessment of patient-reported asthma control. The study has illustrated that this tool has content validity
WHOQOL to assess change | baseline and fourth week
  This questionnaire was represented by the WHO (World Health Organization) and it is used to assess quality and wellbeing of an individual. The study has elaborated the validity and reliability of this tool. Low score on this scale indicates depression and anxiety like symptoms
Oximeter to assess change | baseline and fourth week
  It is an instrument which is used to evaluate oxygen level of blood. This test is performed in various lungs and heart diseases. It is a painless and non-invasive procedure of measuring oxygen saturation. It simply works by placing the device on finger

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Afzal, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Farooq hospital, Khushāb, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andreasson KH, Skou ST, Ulrik CS, Madsen H, Sidenius K, Assing KD, Porsbjerg C, Bloch-Nielsen J, Thomas M, Bodtger U. Breathing Exercises for Patients with Asthma in Specialist Care: A Multicenter Randomized Clinical Trial. Ann Am Thorac Soc. 2022 Sep;19(9):1498-1506. doi: 10.1513/AnnalsATS.202111-1228OC. PMID 35588357
- [Background] Stern J, Pier J, Litonjua AA. Asthma epidemiology and risk factors. Semin Immunopathol. 2020 Feb;42(1):5-15. doi: 10.1007/s00281-020-00785-1. Epub 2020 Feb 4. PMID 32020334
- [Background] Vagedes J, Helmert E, Kuderer S, Vagedes K, Wildhaber J, Andrasik F. The Buteyko breathing technique in children with asthma: a randomized controlled pilot study. Complement Ther Med. 2021 Jan;56:102582. doi: 10.1016/j.ctim.2020.102582. Epub 2020 Oct 23. PMID 33197659
- [Background] Coulson E, Carpenter LM, Georgia TE, Baptist AP. Breathing exercises in older adults with asthma: a blinded, randomized, placebo-controlled trial. J Asthma. 2022 Jul;59(7):1438-1444. doi: 10.1080/02770903.2021.1936015. Epub 2021 Jun 14. PMID 34044738
- [Background] Das RR, Sankar J, Kabra SK. Role of Breathing Exercises in Asthma-Yoga and Pranayama. Indian J Pediatr. 2022 Feb;89(2):174-180. doi: 10.1007/s12098-021-03998-w. Epub 2021 Nov 23. PMID 34812995